CLINICAL TRIAL: NCT04128748
Title: A Phase I/II Study of Liposomal Cytarabine and Daunorubicin (CPX-351) in Combination With Quizartinib in Patients With Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Liposomal Cytarabine and Daunorubicin (CPX-351) and Quizartinib for the Treatment of Acute Myeloid Leukemia and High Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0351; NCI-2019-06051 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0351 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-10-04; First posted 2019-10-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Blasts More Than 10 Percent of Bone Marrow Nucleated Cells; High Risk Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — CPX-351; Injections; Cytarabine; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPX-351, quizartinib) (Experimental): INDUCTION: Patients receive CPX-351 IV over 90 minutes on days 1, 3 and 5 and quizartinib PO on days 6-19. Patients who do not respond to treatment during cycle 1 receive CPX-351 IV on days 1 and 3 and quixartinib PO on days 6-19 during cycle 2. Treatment repeats every 28 days for up 2 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive CPX-351 over 90 minutes on days 1 and 3 and quizartinib PO on days 4-28 of cycle 1. Treatment with CPX-351 repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive quizartinib PO on days 1-28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Drug: Quizartinib

INTERVENTIONS:
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
Drug: Quizartinib — Given PO
  Other Names: AC-220; AC010220; AC220

SUMMARY:
This phase I/II trial studies the side effects and best dose of CPX-351 in combination with quizartinib for the treatment of acute myeloid leukemia and high risk myelodysplastic syndrome. CPX-351, composed of chemotherapy drugs daunorubicin and cytarabine, works in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Quizartinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. The goal of this study is to learn if the combination of CPX-351 and quizartinib can help to control acute myeloid leukemia and myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximum tolerable dose (MTD) of liposomal cytarabine and daunorubicin (CPX-351) in combination with quizartinib in patients with newly diagnosed or relapsed refractory acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (HR-MDS).

II. To determine the overall response rate (ORR) rate including CR (complete remission) + CRp (complete remission with incomplete platelet recovery) + CRi (complete remission with incomplete count recovery) + partial remission (PR) within 3 months of treatment initiation of CPX-351 and quizartinib combination.

SECONDARY OBJECTIVE:

I. To assess the overall survival (OS), event-free survival (EFS) and duration of response (DOR) of patients treated with this combination.

EXPLORATORY OBJECTIVES:

I. To evaluate the ORR, EFS (event free survival) and OS (overall survival) in FLT3 mutated/NPM1 wild-type patients versus FLT3 mutated/NPM1 mutated versus FLT3 wild-type/NPM1 mutated patients treated with CPX-351 and quizartinib.

II. Quantitative changes of FLT3-ITD allelic burden and longitudinal evaluation to identify emergence of FLT3 non-ITD mutations with time in patients treated with the combination.

III. To determine the effect of this treatment combination on responding patients transitioning to hematopoietic stem cell transplant (HSCT).

IV. To store and/or analyze surplus blood or tissue including bone marrow, if available, for potential future exploratory research into factors that may influence development of AML and/or response to the combination (where response is defined broadly to include efficacy, tolerability or safety).

OUTLINE: This is a dose-escalation study of CPX-351, followed by a phase II study.

INDUCTION: Patients receive CPX-351 intravenously (IV) over 90 minutes on days 1, 3 and 5 and quizartinib orally (PO) on days 6-19. Patients who do not respond to treatment during cycle 1 receive CPX-351 IV on days 1 and 3 and quixartinib PO on days 6-19 during cycle 2. Treatment repeats every 28 days for up 2 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive CPX-351 over 90 minutes on days 1 and 3 and quizartinib PO on days 4-28 of cycle 1. Treatment with CPX-351 repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive quizartinib PO on days 1-28 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1) AML (World Health Organization [WHO] classification definition of >= 20% blasts, excluding acute promyelocytic leukemia [APL]), or 2) high risk MDS (> 10% bone marrow blasts)
* For frontline cohort: Patients aged >= 60 years old
* For relapsed or refractory cohort: Patients aged >= 18 years old
* For frontline cohort: Patients must be chemonaive, i.e., not have received any chemotherapy (except hydrea or 1-2 doses of ara-C for transient control of hyperleukocytosis) for AML or MDS. They may have received transfusions, hematopoietic growth factors or vitamins for an antecedent hematological disorder (AHD) or for AML. Temporary prior measures such as apheresis, ATRA (all-trans retinoic acid), steroids or hydrea while diagnostic work-up is being performed are allowed and not counted as a prior salvage. Supportive care therapy for MDS (growth factors, transfusions) will not be considered as prior therapy for MDS/AML and these patients will be enrolled to the frontline cohort of the study if they are otherwise eligible
* For relapsed or refractory cohort: Patients who have received at least one prior therapy for AML or for MDS (with > 10%) blasts will be eligible. Patients may have received up to 4 salvage regimens for AML and/or MDS (defined by the International Prognostic Scoring System [IPSS] classification). Patients who receive MDS directed therapies considered not purely supportive such as hypomethylating agents (HMAs), lenalidomide, investigational therapies, will be enrolled to the salvage cohort if they are otherwise eligible
* In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of protocol therapy will be at least 2 weeks for cytotoxic agents or at least 5 half-lives for cytotoxic/noncytotoxic agents (whichever is shorter). The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochure's, or drug-administration manuals) and will be documented in the protocol eligibility document. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions: (1) intrathecal (IT) therapy for patients with controlled central nervous system (CNS) leukemia at the discretion of the principal investigator (PI). (2) Use of cytarabine (up to 2 g/m^2) or hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy. These medications will be recorded in the case-report form
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Serum biochemical values with the following limits unless considered due to leukemia
* Creatinine < 1.8 mg/dl
* Total bilirubin < 1.8 mg/dL, unless increase is due to hemolysis or congenital disorder
* Transaminases (serum glutamate pyruvate transaminase [SGPT]) < 2.5x upper limit of normal (ULN)
* Potassium, magnesium, and calcium (normalized for albumin) levels should be within institutional normal limits
* Ability to take oral medication
* Ability to understand and provide signed informed consent
* Baseline left ventricular ejection fraction by echocardiogram (ECHO) or multigated acquisition scan (MUGA) >= 50%
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential
* WOCBP must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy until at 30 days after the last dose of investigational drug. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as men with azoospermia do not require contraception. Appropriate methods of birth control include: birth control pills, condoms, intrauterine device (IUD), or other Food and Drug Administration (FDA) approved birth control methods
* Patients may be concurrently enrolling in supportive care clinical trials. Other investigational agents that are used for treatment of other cancers will not be allowed

Exclusion Criteria:

* Patients with known allergy or hypersensitivity to quizartinib, mannitol, CPX-351 or any of their components
* Patients with electrolyte abnormalities at study entry defined as follows: (a) Serum potassium < 3.5 mEq/L despite supplementation, or > 5.5 mEq/L. (b) Serum magnesium above or below the institutional normal limit despite adequate management. (c) Serum calcium (corrected for albumin levels) above or below institutional normal limit despite adequate management
* Patients with known significant impairment of gastrointestinal (GI) function or GI disease as determined by the investigator that may significantly alter the absorption of quizartinib
* Patients with any other known concurrent severe and/or uncontrolled medical condition including but not limited to diabetes, cardiovascular disease including hypertension, renal disease, or active uncontrolled infection, which as determined by the investigator could compromise participation in the study. Patients on active antineoplastic or radiation therapy for a concurrent malignancy at the time of screening. Maintenance therapy, hormonal therapy, or steroid therapy for well-controlled malignancy is allowed
* Patients with a known human immunodeficiency virus (HIV) infection (HIV testing is not required prior to enrollment)
* Patients with known positive hepatitis B or C infection by serology, with the exception of those with an undetectable viral load within 3 months. (Hepatitis B or C testing is not required prior to study entry). Subjects with serologic evidence of prior vaccination to hepatitis B virus (HBV) (i.e., hepatitis surface antigen [HBs Ag]-, and anti-HBs+) may participate
* Patients who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) within 3 days prior to the initiation of study treatment
* Patients who have had any major surgical procedure within 14 days of day 1
* Impaired cardiac function including any of the following: (a) screening electrocardiogram (ECG) with a corrected QT (QTc) > 450 msec. The QTc interval will be calculated by Fridericia's correction factor (QTcF) at screening and on day 6 prior to the first dose of quizartinib. The QTcF will be derived from the average QTcF in triplicate. If QTcF > 450 msec on day 6, quizartinib will not be given
* Patients with congenital long QT syndrome
* History or presence of sustained ventricular tachycardia requiring medical intervention
* Any history of clinically significant ventricular fibrillation or torsades de pointes
* Known history of second or third degree heart block (may be eligible if the patient currently has a pacemaker)
* Sustained heart rate of < 50/minute on pre-entry ECG
* Right bundle branch block + left anterior hemiblock (bifascicular block)
* Complete left bundle branch block
* Patients with myocardial infarction or unstable angina within 6 months prior to starting study drug
* Congestive heart failure (CHF) New York (NY) Heart Association class III or IV
* Atrial fibrillation documented within 2 weeks prior to first dose of study drug
* Patients who are actively taking a strong CYP3A4 inducing medication
* Patients who require treatment with concomitant drugs that prolong QT/QTc interval with the exception of antibiotics, antifungals, and antivirals that are used as standard of care to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the subject or if the Investigator believes that beginning therapy with a potentially QTc-prolonging medication (such as anti-emetic) is vital to an individual subject's care while on study
* Known family history of congenital long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 28 days
  Will follow standard reporting guidelines for adverse events, and summarize safety data by category, severity and frequency.
Complete remission (CRc) rate | Up to 3 cycles (28 days in 1 cycle)
  CRc and toxicity will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey (1995) as extended by Thall and Sung (1998). Will estimate the CRc rate for the combination treatment, along with the 95% credible interval.

SECONDARY OUTCOMES:
Duration of response (DOR) | From the first documentation of CRc to disease recurrence, disease progression or death whichever occurs first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Comparisons of time-to-event endpoint by important covariate subgroups will be made using the log-rank tests.
Event-free survival | From the date of treatment initiation to the date of documented treatment failure, relapses from CRc, or death from any cause,, whichever occurs first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Comparisons of time-to-event endpoint by important covariate subgroups will be made using the log-rank tests.
Overall survival | From treatment start till death or last follow-up id the patients is alive, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Comparisons of time-to-event endpoint by important covariate subgroups will be made using the log-rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Yilmaz, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jentzsch M, Grimm J, Bill M, Brauer D, Backhaus D, Goldmann K, Schulz J, Niederwieser D, Platzbecker U, Schwind S. ELN risk stratification and outcomes in secondary and therapy-related AML patients consolidated with allogeneic stem cell transplantation. Bone Marrow Transplant. 2021 Apr;56(4):936-945. doi: 10.1038/s41409-020-01129-1. Epub 2020 Nov 19. PMID 33208914
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org